CLINICAL TRIAL: NCT01974154
Title: COPD Metabolome, Smoking Oxidants and Aberrant Ciliated Cell Function
Status: Terminated | Type: Observational
Why Stopped: Lack of funding.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1305013966; RFA-HL-12-009 (Other Grant/Funding Number: National Institutes of Health)
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: COPD; Smoking
Keywords: COPD; Smoking; Non-smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung epithelial lining fluid (ELF) obtained by bronchoalveolar lavage (BAL)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort I: A. Healthy nonsmokers B. Healthy smokers C. Healthy smokers/quit smoking D. COPD smokers E. COPD smokers/ quit smoking
  Interventions: Other: Cohort I
- Cohort II: A. Smokers with normal spirometry and normal DLCO B. Smokers, normal spirometry, low DLCO
  Interventions: Other: Cohort II

INTERVENTIONS:
Other: Cohort I — We will evaluate serum and lung ELF obtained by bronchoalveolar lavage, under previous protocols, from 159 individuals at baseline and at 0, 3, 6 and 12 months.
  Groups: Cohort I
Other: Cohort II — Quantify the cilia length on prepared slides from 67 cohort II samples of airway epithelium from biological samples were already obtained from subjects who were consented to participate in prior WCMC IRB approved protocols.
  Groups: Cohort II

SUMMARY:
Cigarette smoking is the major cause of chronic obstructive pulmonary disease (COPD), the 4th cause of mortality in the US. Central to COPD pathogenesis is "ciliopathy", dysfunction of the airway ciliated cells that mediate transport of mucus to remove inhaled pathogens. The focus of this study is to carry out metabolic profiling of banked biologic samples and assess the hypothesis that COPD is associated with a unique metabolome in serum and lung epithelial lining fluid, and that subsets of the COPD metabolome are linked to the ciliopathy of COPD.

DETAILED DESCRIPTION:
Cigarette smoking is the major cause of chronic obstructive pulmonary disease (COPD), the 4th cause of mortality in the US. Central to COPD pathogenesis is "ciliopathy", dysfunction of the airway ciliated cells that mediate transport of mucus to remove inhaled pathogens. The COPD ciliopathy leads to mucus accumulation, impaired host defense and recurrent infections. Using a state-of-the-art platform for global metabolite profiling and unique cohorts with serum and lung biologic samples, our deliverables are to identify a metabolome focused on biomarkers related to airway ciliopathy in COPD, and use the observed metabolic changes to: (1) direct mechanistic studies to define ciliopathy at a molecular level; (2) identify novel targets for therapeutic intervention in COPD; and (3) identify smokers at high risk for COPD. Preliminary metabolic data led to our first clues - COPD smokers have decreased serum citrulline levels, consistent with a deficiency in lung nitric oxide synthase (NOS) activity, and thus lung nitric oxide (NO) deficiency. This, together with supporting data of a smoking-induced NOS/NO-related ciliopathy, and knowledge that smokers have significant oxidant-related changes in the airway epithelial transcriptome, led to our aims, combining metabolomics of defined cohorts, murine and human mechanistic studies and computational / statistical integration.

Aim 1. To carry out metabolic profiling of banked biologic samples of our characterized cohorts to assess the hypothesis that COPD is associated with a unique metabolome in serum and lung epithelial lining fluid, and that subsets of the COPD metabolome are linked to the ciliopathy of COPD.

Aim 2. To combine metabolic profiling and in vitro studies of human and murine airway epithelium to evaluate the hypothesis that there is a link between the COPD metabolome (focusing on the inferred NO deficiency) and mechanisms underlying the ciliopathy of COPD.

Aim 3. Characterize and quantify the cigarette smoke induced "redoxome" in lung and serum and assess its role in ciliated cell dysfunction. Studies seek to identify a link between smoking, a burden of oxidants to the lung epithelium and the pathogenesis of COPD - potentially providing biomarker(s) that predict which smokers will develop COPD and identifying new targets for therapy of COPD.

ELIGIBILITY:
Inclusion Criteria:

All study subjects should be able to provide informed consent Males or females ages 18 years and older Must provide HIV informed consent Lung disease proven by at least one of the following: symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and/or (6) diseases of organs with known association with lung disease

Exclusion Criteria:

Individuals not deemed in good overall health by the investigator will not be accepted into the study.

Habitual use of drugs and/or alcohol within the past six months (Acceptable: Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria).

Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.

Individuals with allergies to atropine or any local anesthetic will not be accepted into the study.

Individuals with allergies to pilocarpine, isoproterenol, terbutaline, atropine or aminophylline will not be accepted into the study.

Females who are pregnant or nursing will not be accepted into the study Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic will not be included in the study Patient refuses consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Gene expression changes in airway epithelium | One year
  We will perform metabolic profiling of biologic samples to assess the hypothesis that smoking-induced COPD is associated with a unique metabolome in serum and lung ELF, and that subsets of the COPD metabolome are linked to the ciliopathy of COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College - Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided